CLINICAL TRIAL: NCT01674907
Title: Non-interventional Study of Avastin in 1st Line Metastatic Colorectal Cancer
Brief Title: An Observational Study of Avastin (Bevacizumab) in First Line in Patients With Metastatic Colorectal Cancer (AVANiS)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22399
Record Dates: First submitted 2012-08-22; First posted 2012-08-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the use in clinical practice and the efficacy of Avastin (bevacizumab) in patients with metastatic colorectal cancer who have not received prior chemotherapy treatment in the metastatic setting. Patients for whom the treating physician has decided to initiate therapy with Avastin will be followed for 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically confirmed metastatic colorectal cancer without prior chemotherapy in the metastatic setting

Exclusion Criteria:

* Contraindications for Avastin according to the locally approved package insert (version 7 April 2006)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer without prior chemotherapy in the metastatic setting
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Dosage/schedule of 1st-line Avastin | approximately 3 years
Duration of treatment | approximately 3 years
Chemotherapy regimens used in clinical practice | approximately 3 years
Clinical/demographic patient characteristics at baseline | approximately 3 years

SECONDARY OUTCOMES:
Progression-free survival | approximately 3 years
Relationship between termination of Avastin treatment and time point of progression | approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- South Africa (5):
  - Cape Town
  - George
  - Port Elizabeth
  - Pretoria
  - Vereeniging